CLINICAL TRIAL: NCT06203821
Title: A Pilot Study of Perioperative NP137 and FOLFIRINOX in Resectable Pancreatic Cancer
Brief Title: Study of Perioperative NP137 and FOLFIRINOX in Resectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aram Hezel (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor-Investigator, Aram Hezel, Professor, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMGIP25077
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; FOLFIRINOX; NP137; Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — netrin-1 inhibitor NP137

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patient receive two doses of the study drug, NP137, approximately two weeks apart. This will be followed by surgery. After the surgery if feasible, patients will begin post-surgical treatment with a standard-of-care chemotherapy regimen called FOLFIRINOX, combined with the study drug, NP137, for a total duration of about 6 months. Upon completing this phase, patients will receive an additional 6 months of treatment with only the study drug NP137.
  Interventions: Drug: NP137

INTERVENTIONS:
Drug: NP137 — NP137 for the Treatment of Resectable Pancreatic Cancer

SUMMARY:
The objective of this study is to investigate whether adding the study drug, NP137, to a patient's treatment regimen (before surgery and in combination with chemotherapy afterward) can alter the behavior of pancreatic cancer..

DETAILED DESCRIPTION:
The aim of this study is to evaluate the mechanism of action for a novel anti-Netrin-1 antibody (NP137) in patients with pancreatic ductal adenocarcinoma. Pre-clinical data indicates that anti-Netrin-1 therapy can prevent/delay metastatic progression of disease by inducing cancer cell death through its dependence receptor Unc5b as well as prevent epithelial to mesenchymal transition (EMT).

This pilot study is designed to provide vital translational scientific information that will inform the design of future clinical trials for NP137. This information includes determining the optimal use of NP137 with cytotoxic, as well as the treatment setting of resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with imaging suggesting resectable pancreatic cancer and without strong evidence of metastatic disease.
* Accept to undergo biopsy for initial diagnosis and research purposes. NOTE: For patients who already have cytologically or histologically confirmed resectable pancreatic ductal adenocarcinoma, they must agree to undergo research biopsy.
* Cytologically or histologically confirmed resectable pancreatic ductal adenocarcinoma.
* Confirmed resectable pancreatic ductal adenocarcinoma by treating surgeon.
* No prior systemic therapy, radiation therapy, or resection for pancreatic cancer.
* Written informed consent to participate in the trial.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 and ability to undergo perioperative systemic therapy, radiation therapy and surgery as deemed by the treating investigator.
* Adequate bone marrow and organ function
* Subjects of childbearing potential must have a negative urine or serum pregnancy test prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required for enrollment.
* Subjects of child-bearing potential must agree to use adequate contraception E.g. hormonal , barrier method of birth control, and abstinence prior to study entry, for the duration of study treatment, and for 6 months after completion of study therapy. Subject who become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform their treating physician immediately. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study therapy, subjects should agree to discontinue breastfeeding prior enrollment in the study.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand a written informed consent document, and ability and willingness to comply with study procedures for the entire length of the study. Patients with impaired decision-making capacity (IDMC) who have a close caregiver or legally authorized representative (LAR) and/or family member who can make may decision on the patient behalf may enroll in the trial per the enrolling physician assessment.

Exclusion Criteria:

* Patients with borderline or locally advanced or metastatic pancreatic cancer as deemed by treating surgeon.
* Patients who are unlikely to undergo surgery, and systemic therapy, in the opinion of the treating investigators.
* Patients with grade ≥ 2 peripheral neuropathy.
* Patients with known Gilbert's Syndrome, Dihydropyrimidine dehydrogenase (DPD) deficiency, or homozygosity for UGAT1A1*28 polymorphism. Note: evaluation for these is not required.
* Patients with active duodenal or gastric ulcers, or direct tumor invasion of the bowel or stomach by endoscopic evaluation. Note: patients with previous ulcers without active bleeding or symptoms are eligible.
* Patients with serious active infection within 2 weeks prior to enrollment (e.g. requiring hospitalization and/or intravenous [IV] antibiotics) or currently receiving oral or IV antibiotics for the treatment of infection. Patients receiving prophylactic antibiotics are eligible.
* Patients with known untreated hepatitis B or C (HBV/HCV) or known human immunodeficiency virus (HIV). Note: evaluation for these is not required.
* Patients with uncontrolled intercurrent illness within 3 months prior to start of study treatment that could substantially increase risk of incurring AEs in the opinion of the treating investigator, including but not limited to:

  * Uncontrolled hypertension, despite optimal medical management, hypertensive crisis, or hypertensive encephalopathy,
  * Symptomatic congestive heart failure [CHF],
  * Uncontrolled cardiac arrhythmia, or
  * Current psychiatric illness/social situations or other conditions that would limit compliance with study requirements or.
* Patients with known concurrent malignancy that is expected to require active treatment within two years or may interfere with the interpretation of the efficacy and safety outcomes of this study in the opinion of the treating investigator. Note: Superficial bladder cancer, nonmelanoma skin cancers, and low-grade prostate cancer not requiring cytotoxic therapy should not exclude participation in this trial. Patients with CLL may be enrolled if they do not require active chemotherapy and their hematologic, renal and hepatic function meets criteria previously mentioned.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications in the opinion of the treating investigator.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Determining if NP137 can shift the primary tumor MAK's Signature Epithelial-to-Mesenchymal Transition (EMT) Mean Score towards a more epithelial phenotype | 3-5 years
  EMT score is determined by the mean expression of mesenchymal genes minus the mean expression of epithelial genes Therefore, a positive EMT score suggests a mesenchymal status (worse outcome), whereas a negative score indicates an epithelial status (better outcome).

SECONDARY OUTCOMES:
Pathological Response Rate | 3-5 years
  Pathologic response rate after treatment with NP137. The Pathological Response definition will follow the College of American Pathologists criteria
Two-year metastasis-free survival | 4-7 years
  Metastasis-free survival at two years. Metastasis-free survival is defined as the time between the date of enrollment and the date of the 1st distant event occurrence .
Disease free survival | 5-8 years
  Disease free survival defined as time from the date of enrollment until the date of the first cancer-related event, second cancer, or death from any cause.
Overall survival | 5-8 years
  Overall survival is defined by the date of enrollment to date of death from any cause
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 5-8 years
  Descriptive of Adverse event during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Aram Hezel, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No